CLINICAL TRIAL: NCT04194528
Title: Feasibility of a Digital Medicine Program in Optimizing Opioid Pain Control in Cancer Patients
Brief Title: S1916 Digital Medicine Program for Pain Control in Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study sponsor withdrew support.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: Proteus Digital Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S1916
Record Dates: First submitted 2019-12-06; First posted 2019-12-11 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Oxycodone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Oxycodone/acetaminophen (5/325 mg) DMP (Experimental): The intervention is the Proteus digital medicine program consisting of a mobile application, a patch worn on the body, and oxycodone/acetaminophen 5/325 mg co-encapsulated with ingestible sensors. The duration of the intervention is 6 weeks.
  Interventions: Drug: Oxycodone/acetaminophen 5/325 mg; Device: Proteus digital medicine program

INTERVENTIONS:
Drug: Oxycodone/acetaminophen 5/325 mg — The intervention is the Proteus digital medicine program consisting of a mobile application, a patch worn on the body, and oxycodone/acetaminophen 5/325 mg co-encapsulated with ingestible sensors. The duration of the intervention is 6 weeks.
Device: Proteus digital medicine program — The intervention is the Proteus digital medicine program consisting of a mobile application, a patch worn on the body, and oxycodone/acetaminophen 5/325 mg co-encapsulated with ingestible sensors. The duration of the intervention is 6 weeks.

SUMMARY:
This is a feasibility study to assess the use of a Digital Medicine Program (consisting of an FDA-approved ingestible sensor co-encapsulated with oxycodone/acetaminophen (5 mg/325 mg), a small wearable patch, and a mobile application) in cancer patients with metastatic disease experiencing uncontrolled pain.

DETAILED DESCRIPTION:
Given the high prevalence of cancer pain and issues with undertreatment and opioid misuse, focused efforts to improve monitoring of medication ingestion patterns are needed. This study will test the feasibility of using a Digital Medicine Program (consisting of an FDA-approved ingestible sensor co-encapsulated with oxycodone/acetaminophen (5 mg/325 mg), a small wearable patch, and a mobile application) in cancer patients with metastatic disease experiencing uncontrolled pain. Data collected from this study (such as information on patterns of DMP usage by patients and physicians and changes to medication dosage based on the reported symptoms) will inform the design of a randomized controlled trial of the DMP vs. usual care to control cancer pain and increase quality of life. If successful, this DMP could be a new way for physicians to evaluate patients' pain medication use patterns and titrate for adequate pain control while concurrently monitoring for adverse effects or abusive/addictive behavior. It will also promote improved communication between patients and their physicians and potentially address and ease some of patients' concerns and hesitancies regarding opioid medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic cancer
* Patients must have a worst pain score of at least 3 (on a scale of 0-10) on the Brief Pain Inventory (BPI)* within 3 days prior to registration and be deemed by their physician to require initiation, continuation, or uptitration of opioid therapy with oxycodone/acetaminophen 5mg/325mg.
* Patients currently on oxycodone/acetaminophen are eligible as long as they are on the 5 mg/325 mg dose.
* Patients currently on another opiate, who have been prescribed or will be prescribed oxycodone/acetaminophen as an addition to their therapy are also eligible.
* Patients must be >/= 18 years of age
* Patients must complete the baseline PRO questionnaires prior to registration.
* Patients must be able to read English, as the ePRO questionnaires are in English and patient instructions on the Proteus Discover mobile application are in English.
* Patients must be willing to participate in electronic data collection and must have an iPhone, Android phone, or tablet with cellular connectivity in order to download the Patient Cloud and Proteus Discover mobile applications onto his/her device.
* Patients must have successfully downloaded the Proteus Discover App.
* Patients must not have a known allergy to adhesive tape, hydrogel or conductive gel, or hydrocolloid. (The adhesive strip for the Wearable Sensor Patch does not contain natural latex rubber).
* Patients of reproductive potential must have agreed to use an effective contraceptive method. All men are considered to be of reproductive potential unless they have had a vasectomy or orchiectomy.

Exclusion Criteria:

* Women must not be pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, M.D., M.S., Study Chair — SWOG Cancer Research Network
Locations (5):
- United States (5):
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Cancer Center NCORP, Urbana, Illinois
  - Montana Cancer Consortium, Billings, Montana
  - Columbia University, New York, New York
  - PRISMA Health Upstate Cancer Institute, Greenville, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 55.4 [51.8 to 59.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Determined by Accrual, Adherence and Patient Retention.
Description: Feasibility will be determined by accrual (as confirmed by registration to the trial), adherence and patient retention (as measured and relayed by the wearable patch/sensor).
Time Frame: adherence and retention - 6 weeks; accrual - 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Pain Levels and Pain Interference With Daily Activity
Description: Pain levels are measured by average pain score and pain interference with daily activity score at 2, 4, and 6 weeks on the Brief Pain Inventory-Short Form (BPI-SF). Also, pain in the last 24 hours is measured daily using the worst pain item from the BPI-SF. Pain is rated on a scale of 0-10 with 10 signifying the worst symptoms.
Time Frame: 2, 4, and 6 weeks.
Population: Study only accrued 2 patients and had difficulty getting sites to participate in a trial with a controlled substance. Study was ultimately discontinued when the DMP software company went bankrupt and was sold. Due to the lack of patient data, only the primary objective was analyzed.
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

3. Secondary Outcome: Opioid Medication Consumption
Description: Opioid medication consumption is assessed as the number of pills taken over the number of study pills prescribed.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

4. Secondary Outcome: Unplanned Hospital and Emergency Department Visits
Description: Unplanned hospital and emergency department visits assessed as any reported unplanned visits because of pain between the date of registration and the 6-week follow-up timepoint.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of Changes in Pain Management Regimen
Description: Frequency of changes in pain management regimen is measured as any change in the dosage, frequency, or the pain medication between baseline and 6-week follow-up.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

6. Secondary Outcome: Activity Levels
Description: Activity levels are measured as active time and rest time in minutes and total daily step count.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

7. Secondary Outcome: Patient Somatic Symptoms
Description: Patient somatic symptoms of opioid treatment will be measured using the Edmonton Symptom Assessment (revised version). Questions are rated on a scale of 1-10 with 10 being "worst" outcome.
Time Frame: baseline 2, 4, and 6 weeks.
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

8. Secondary Outcome: Patient Satisfaction With the Digital Medicine Program (DMP).
Description: Patient satisfaction will be assessed by survey that measures patient satisfaction on a scale of 1-5 with the higher score having the better outcome.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

9. Secondary Outcome: Provider Satisfaction With Digital Medicine Program (DMP)
Description: Provider satisfaction will be assessed by survey that measures provider satisfaction on a scale of 1-5 with the higher score having the better outcome.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

10. Secondary Outcome: ePRO Feasibility
Description: ePRO feasibility will be defined by the extent of missing data at each assessment time for those items or instruments required to be completed using the Patient Cloud ePRO app; assessing the patient experience of using the Patient Cloud ePRO app with a one-time questionnaire at the conclusion of the study.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

11. Secondary Outcome: Patient Psychological Distress
Description: Patient depression and anxiety will be measured using the Patient Health Questionnaire (PHQ-4). Questions are rated on a scale of 0-3 with higher score having the worst outcome.
Time Frame: 2, 4, and 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

12. Secondary Outcome: Patient Global Quality of Life
Description: Patient quality of life (including anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, satisfaction with participation in social roles and activities and single pain intensity) will be measured using the PROMIS-29. Patients respond to questions by marking one response: very poor, poor, fair, good and very good.
Time Frame: 2, 4, and 6 weeks
Population: as for outcome 2
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events are monitored and collected at the 2, 4, and 6-week follow up visits.
Description: Patients will complete the S1916 Opioid Adverse Event Survey (See Section 14.4) at the 2, 4, and 6-week follow-up visits to report the frequency with which they experience several potential adverse effects. Sites will collect side effect data at the same interval on the S1916 Adverse Events form and code using CTCAE 5.0. The rare adverse effects associated with the Digital Medicine Program (ingestible sensor and patch) will be collected on S1916 Follow-Up form.
Arm/Group | Oxycodone/Acetaminophen (5/325 mg) DMP
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Acetaminophen (5/325 mg) DMP (N=2)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 2 participants were accrued due to COVID-19 limiting enrollment in sites and the extreme difficulty in getting sites to participate in the trial due to the use of a controlled substance as state regulations varied. The study was discontinued when the company providing the DMP and associated software went bankrupt and was acquired by a company that had no interest in continuing the trial. Due to a lack of patient data, we did not analyze any of objectives other than telemedicine feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT04194528/Prot_SAP_ICF_001.pdf